CLINICAL TRIAL: NCT00711763
Title: Calciuric Effect and Cyclic Parenteral Nutrition in Preterm Infants
Status: Terminated | Type: Observational
Why Stopped: failure to recruit more patients and lack of supporting personnel.
Sponsor: Louisiana State University Health Sciences Center Shreveport (Other)
Responsible Party: Sponsor
Other Study IDs: H08-048
Record Dates: First submitted 2008-07-03; First posted 2008-07-09 (Estimated); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Preterm Infants; Metabolic Bone Disease
Keywords: Preterm Infant; Parenteral nutrition cycling; TPN cycling; Hypercalcuria
MeSH Terms: conditions — Bone Diseases, Metabolic; Premature Birth; Hypercalciuria

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of our work is to study the effect of total parenteral nutrition (TPN) cycling in preterm infants on hypercalcuria (excessive calcium excretion in urine). TPN cycling refers to administering the TPN over a portion of the day rather than the whole day. Our hypothesis is that cyclic TPN includes more hypercalcuria in preterm infants as compared to continuous TPN.

Objectives:

Measure Urinary Calcium(Ca) during the periods of continuous and cyclic TPN.

Compare the amount of Ca losses in the urine continuous vs. cyclic TPN

DETAILED DESCRIPTION:
Randomized cross over design, in which babies will receive TPN either continuously or on a cyclic basis for 3 days. The patients will then be crossed over to receive the other way of administration over the following 3 days, thus each patient will serve as his or her own control. Continuous TPN will be administered over 24 hours for 3 days, while the cyclic TPN will be given for 18 hours then followed by a Dextrose only solution at the same concentration and rate as the TPN for 6 hours. Trophic feeds up to 20 ml/kg/day will be allowed throughout the study period at the discretion of the attending neonatologist.

ELIGIBILITY:
Inclusion Criteria:

* Preterm babies with birth weights of 1500 gm or less.
* Expected to be restricted from oral feeding or on trophic feeds
* On TPN for at least 6 days

Exclusion Criteria:

* Infants who at the time of enrollment are on any diuretics (Lasix, hydrochlorothiazide, Aldactone, etc.) or caffeine
* those who are hemodynamically unstable
* Or have renal or hepatic insufficiency
* Infants with major congenital anomalies

Ages: 1 Hour to 9 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Patients will be recruited from the NICU at (LSUHSC) after obtaining parental consent.
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2008-07; Primary Completion 2011-04 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sameh Hussein, M.D., Principal Investigator — Louisiana State University Health Science Center-Shreveport
Locations (1):
- Louisiana State University Health Science Center-Shreveport, Shreveport, Louisiana, United States

REFERENCES:
- [Background] Hurley DL, McMahon MM. Long-term parenteral nutrition and metabolic bone disease. Endocrinol Metab Clin North Am. 1990 Mar;19(1):113-31. PMID 2113469
- [Background] Koo WW, Tsang RC, Succop P, Krug-Wispe SK, Babcock D, Oestreich AE. Minimal vitamin D and high calcium and phosphorus needs of preterm infants receiving parenteral nutrition. J Pediatr Gastroenterol Nutr. 1989 Feb;8(2):225-33. doi: 10.1097/00005176-198902000-00017. PMID 2496213
- [Background] Koo WW, Sherman R, Succop P, Krug-Wispe S, Tsang RC, Steichen JJ, Crawford AH, Oestreich AE. Fractures and rickets in very low birth weight infants: conservative management and outcome. J Pediatr Orthop. 1989 May-Jun;9(3):326-30. PMID 2723052
- [Background] Ferrone M, Geraci M. A review of the relationship between parenteral nutrition and metabolic bone disease. Nutr Clin Pract. 2007 Jun;22(3):329-39. doi: 10.1177/0115426507022003329. PMID 17507733
- [Background] Shike M, Harrison JE, Sturtridge WC, Tam CS, Bobechko PE, Jones G, Murray TM, Jeejeebhoy KN. Metabolic bone disease in patients receiving long-term total parenteral nutrition. Ann Intern Med. 1980 Mar;92(3):343-50. doi: 10.7326/0003-4819-92-3-343. PMID 6766694
- [Background] Shike M, Shils ME, Heller A, Alcock N, Vigorita V, Brockman R, Holick MF, Lane J, Flombaum C. Bone disease in prolonged parenteral nutrition: osteopenia without mineralization defect. Am J Clin Nutr. 1986 Jul;44(1):89-98. doi: 10.1093/ajcn/44.1.89. PMID 3088971
- [Background] Klein GL, Targoff CM, Ament ME, Sherrard DJ, Bluestone R, Young JH, Norman AW, Coburn JW. Bone disease associated with total parenteral nutrition. Lancet. 1980 Nov 15;2(8203):1041-4. doi: 10.1016/s0140-6736(80)92271-0. PMID 6107676
- [Background] Aladangady N, Coen PG, White MP, Rae MD, Beattie TJ. Urinary excretion of calcium and phosphate in preterm infants. Pediatr Nephrol. 2004 Nov;19(11):1225-31. doi: 10.1007/s00467-004-1574-1. PMID 15349762
- [Background] Atkinson SA, Shah JK, McGee C, Steele BT. Mineral excretion in premature infants receiving various diuretic therapies. J Pediatr. 1988 Sep;113(3):540-5. doi: 10.1016/s0022-3476(88)80648-6. PMID 3411401
- [Background] Pelegano JF, Rowe JC, Carey DE, LaBarre DJ, Edgren KW, Lazar AM, Horak E. Effect of calcium/phosphorus ratio on mineral retention in parenterally fed premature infants. J Pediatr Gastroenterol Nutr. 1991 Apr;12(3):351-5. doi: 10.1097/00005176-199104000-00011. PMID 1649288
- [Background] Linkswiler HM, Zemel MB, Hegsted M, Schuette S. Protein-induced hypercalciuria. Fed Proc. 1981 Jul;40(9):2429-33. PMID 7250387
- [Background] Wood RJ, Bengoa JM, Sitrin MD, Rosenberg IH. Calciuretic effect of cyclic versus continuous total parenteral nutrition. Am J Clin Nutr. 1985 Mar;41(3):614-9. doi: 10.1093/ajcn/41.3.614. PMID 3919560
- [Background] Btaiche IF, Khalidi N. Parenteral nutrition-associated liver complications in children. Pharmacotherapy. 2002 Feb;22(2):188-211. doi: 10.1592/phco.22.3.188.33553. PMID 11837558
- [Background] Collier S, Crough J, Hendricks K, Caballero B. Use of cyclic parenteral nutrition in infants less than 6 months of age. Nutr Clin Pract. 1994 Apr;9(2):65-8. doi: 10.1177/011542659400900265. PMID 8078440
- [Background] Takehara H, Hino M, Kameoka K, Komi N. A new method of total parenteral nutrition for surgical neonates: it is possible that cyclic TPN prevents intrahepatic cholestasis. Tokushima J Exp Med. 1990 Dec;37(3-4):97-102. PMID 2128784